CLINICAL TRIAL: NCT07239440
Title: A Multicenter, Double-blind, Active-controlled, Randomized, Parallel Clinical Trial to Evaluate the Efficacy and Safety of DA-2811 When Added to Ongoing BT-1 and BT-2 Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DA-2811 When Added to Ongoing BT-1 and BT-2 Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA2811_DMLD_II
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA-2811 (Experimental): DA-2811 + DA-2811-R2
  Interventions: Drug: DA-2811
- DA-2811-C (Experimental): DA-2811-C + DA-2811-R1
  Interventions: Drug: DA-2811-C

INTERVENTIONS:
Drug: DA-2811 — DA-2811 + DA-2811-R2, orally, once daily
  Arms: DA-2811
Drug: DA-2811-C — DA-2811-C + DA-2811-R1, orally, once daily
  Arms: DA-2811-C

SUMMARY:
This study is a multicenter, double-blind, active-controlled, randomized, parallel clinical trial to evaluate the efficacy and safety of DA-2811 when added to ongoing BT-1 and BT-2 combination therapy in patients with type 2 diabetes who have inadequate glycemic control

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type II diabetes mellitus aged 19 years or older
2. Patients with fasting plasma glucose≤270mg/dL at the screening visit
3. Patients with 18.5kg/m^2≤BMI≤40kg/m^2 at the screening visit
4. Patients who have signed an informed consent themselves after receiving detailed explanation about the clinical study

Exclusion Criteria:

1. Patients with type 1 diabetes, secondary diabetes, gestational diabetes, diabetic coma or -pre-coma, metabolic acidosis including lactic acidosis and diabetic ketoacidosis
2. Patients with a medical history of New York Heart Association(NYHA) class III~IV heart failure or with congestive heart failure, acute and unstable heart failure
3. Patients with severe infectious disease or severe traumatic systemic disorders
4. Patients with hypopituitarism or adrenal insufficiency, pulmonary infarction, severe pulmonary dysfunction and other hypoxemia
5. Patients with galactose intolerance, lapp lactase deficiency, glucosegalactose malabsorption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Change from baseline at 12 weeks

SECONDARY OUTCOMES:
HbA1c | Change from baseline at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea